CLINICAL TRIAL: NCT02304198
Title: A Single-arm, Open-label, Extension Study to Evaluate the Long-term Safety of Udenafil in Patient With Pulmonary Arterial Hypertension(PAH)
Brief Title: Clinical Trial to Evaluate the Long-term Safety of Udenafil in Patient With PAH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA8159_PAH_EX
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Udenafil (Experimental): Udenafil 50mg tablet by mouth, every 12 hours for 1-year(48-weeks)
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — Udenafil 50mg tablet
  Other Names: Zydena

SUMMARY:
This study evaluates the long-term safety of Udenafil in Patient with Pulmonary Arterial Hypertension(PAH). All the patients will receive Udenafil for 1-year(48-weeks).

DETAILED DESCRIPTION:
Pulmonary arterial Hypertension is characterized by a progressive incerease in pulmonary vascular resistance(PVR) leading to right ventricualar failure.

Udenafil inhibits PDE 5, an enzyme that metabolizes cGMP, enhancing the cGMP mediated relaxation and growth inhibition of vascular smooth muscle cells, including those in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the initial study(DA8159_PAH_II), 12-week, double-blind, placebo-controlled trial

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse Events, Physical Examination, Vital Sign, Electrocardiography, Laboratory test, etc) | during 48-weeks
  Adverse Events, Physical Examination, Vital Sign, Electrocardiography, Laboratory test, etc

SECONDARY OUTCOMES:
6-MWD | 24, 48-week
BORG dyspnea score | 24, 48-week
WHO class | 12, 24, 36, 48-week
Time to clinical worsening(TTCW) | during 48-weeks
NT-pro BNP | 24, 48-week
Echocardiography | 48-week

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Kyung Kim, M.D., Ph.D., Study Chair — Samsung Medical Center; Sung-A Jang, M.D., Ph.D., Principal Investigator — Samsung Medical Center; Jun-Bin Park, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Hyung-Kwan Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Hyuk-Jae Jang, M.D., Ph.D., Principal Investigator — Severance Hospital; Hae-Ok Jung, M.D., Ph.D., Principal Investigator — Seoul St. Mary's Hospital; Jung-Hyun Choi, M.D., Ph.D., Principal Investigator — Pusan National University Hospital; Jae-Seung Lee, M.D., Ph.D., Principal Investigator — Asan Medical Center; Kye-Hun Kim, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Jin-Ok Jeong, M.D., Ph.D., Principal Investigator — Chungnam National University Hospital; Sang-Yeub Lee, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, Irwon-Dong 50, South Korea